CLINICAL TRIAL: NCT01434927
Title: Unsedated Colonoscopy: An Option For Some But Not For All
Brief Title: The Clinical Acceptability of Unsedated Colonoscopy
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Principal Investigator, MD, Valduce Hospital
Other Study IDs: 07CE2009
Record Dates: First submitted 2011-08-18; First posted 2011-09-15 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colonoscopy outpatients: All patients referred to our Unit to undergo colonoscopy for any indication
  Interventions: Procedure: Unsedated colonoscopy

INTERVENTIONS:
Procedure: Unsedated colonoscopy — Patients were offered to undergo colonoscopy without routine premedication
Procedure: Unsedated colonoscopy — Patients were offered to undergo unsedated procedure. Their demographics and clinical data were recorded

SUMMARY:
The study was aimed to prospectively evaluate the acceptance rate of unsedated colonoscopy, in a setting where routine sedation for colonoscopy is standard practice and to characterize the subset of patients willing to try and potentially completing an unsedated procedure.

DETAILED DESCRIPTION:
Patients were offered to undergo colonoscopy without routine premedication. In case of both acceptance and refusal, a brief questionnaire recording demographics (gender, age, level of education) and clinical features was prospectively recorded in a standard data sheet by one of the four endoscopists at enrollment. Clinical features recorded for each patient included: indication to the procedure, history of abdominal surgery or irritable bowel syndrome, presence of pain as main symptom, chronic use of sedative medications, level of patient's anxiety (none, mild, moderate or severe), main concern about the examination and reason for willing to attempt unsedated procedure.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients

Exclusion Criteria:

1. previous colorectal surgery
2. indication to a bi-directional endoscopy
3. indication to a partial examination
4. patients' refusal or inability to provide informed consent and
5. advanced heart, lung, liver or renal disease (American Society of Anesthesiology risk class III-IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive 18-80 year-old outpatients presenting to undergo open-access colonoscopy for routine indications were considered eligible to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
ODDS ratio for unsedated colonoscopy acceptance | up to 8 months
  Multivariate analysis was used to assess the association of dempgraphics (gender, age, level of education) and clinical features (indication to the procedure, history of abdominal surgery or irritable bowel syndrome, presence of pain as main symptom, chronic use of sedative medications, level of patient's anxiety (none, mild, moderate or severe), main concern about the examination and reason for willing to attempt unsedated procedure) to the acceptance of unsedated colonoscopy

SECONDARY OUTCOMES:
Acceptance rate of unsedated colonoscopy | up to 8 months
  Proportion of patients accepting to attempt colonoscopy without routine premedication
ODDS ratios for unsedated colonoscopy completion | up to 8 months
  Multivariate analysis was used to assess the association of dempgraphics (gender, age, level of education) and clinical features (indication to the procedure, history of abdominal surgery or irritable bowel syndrome, presence of pain as main symptom, chronic use of sedative medications, level of patient's anxiety (none, mild, moderate or severe), main concern about the examination and reason for willing to attempt unsedated procedure) to the completion of unsedated colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Franco Radaelli, MD, Principal Investigator — Valduce Hospital
Locations (1):
- Vadluce Hospital, Como, Italy